CLINICAL TRIAL: NCT02545634
Title: Effects of a Probiotic Supplement on Symptoms of ADHD and Anxiety in Children
Brief Title: Effects of a Probiotic Supplement on Symptoms of Attention Deficit Hyperactivity Disorder and Anxiety in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acadia University (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: APB-C1
Record Dates: First submitted 2015-07-30; First posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Attention Deficit Hyperactivity Disorder; Anxiety
Keywords: probiotic; ADHD; anxiety; digestive health; children; attention deficit; gut brain axis; nutritional supplement; microbiome
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo powder (Placebo Comparator): Placebo powder contains the same ingredients as the probiotic powder except the L. helveticus R0052 and B. longum R0175. All participants will consume the placebo for 28 days during one of two dosing phases.
  Interventions: Other: Placebo
- Probiotic powder (Experimental): The Investigational Product is formulated with a combination of two active ingredients: L. helveticus R0052 and B. longum R0175 and the percentage of each strain is 90% and 10% respectively. The minimum total count of L. helveticus R0052 and B. longum R0175 is 3 x 109 colony forming units (CFU) per stick during the shelf-life. The IP also contains the following excipients: xylitol (sweetener), maltodextrin (coating agent), fruit flavor and malic acid (acidity regulator). The total weight is 1.5 g per stick. All participants will consume the placebo for 28 days during one of two dosing phases.
  Interventions: Dietary Supplement: L. helveticus R0052 and B. longum R0175

INTERVENTIONS:
Dietary Supplement: L. helveticus R0052 and B. longum R0175 — See arm descriptions for intervention description.
  Other Names: Probiostick; Jamieson Probiotic Sticks; Health Canada Natural Product Number (NPN) 80021343
  Arms: Probiotic powder
Other: Placebo
  Arms: Placebo powder

SUMMARY:
The study will examine the effect of a probiotic supplement (Lactobacillus helveticus R0052 and Bifidobacterium Longum R0175) dissolved in a dairy product such as milk or ice-cream on symptoms of ADHD and anxiety in children. The main goal is to determine if probiotics might be useful as a treatment for anxiety and ADHD symptoms in children. A second goal is to examine the effects of probiotics on saliva cortisol levels. Finally, the investigators are also interested in the effects of the probiotics on children's digestive health.

DETAILED DESCRIPTION:
Participants will be recruited using information distributed through schools in the Annapolis Valley area and with the use of advertising campaigns visible across Nova Scotia as previously described. Interested participants will be directed to the study's website (www.probioticstudy.com), where they will be able to view a complete summary of the study's timeline and details. After reviewing the website, guardians of potential participants will be able to complete an initial consent form and preliminary questionnaire in order to determine their child's eligibility for participation. The process of completing the consent form and initial questionnaires is expected to take approximately 15 minutes. Participants' responses to the preliminary questionnaire will be reviewed by the researchers, and initial appointments will be scheduled, either at the Acadia University location or the Halifax location.

Each participant will be enrolled in the study for a thirteen-week period with a six-month follow-up session. The first week will be an information-gathering week during which participants will complete a daily food diary online with their parents' assistance. Each evening during this initial week, and at the end of each week throughout the study period, the child will answer a few questions about his or her symptoms of anxiety and/or ADHD, and gastrointestinal health. Parents/guardians will answer parallel questions about the child's symptoms of anxiety and/or ADHD.

Confidentiality will be maintained by assigning each participant a code number based on the last four digits of their phone number and the first letter of their last name when they begin the study (for siblings the first letter of their first name will be used). The food diary and all other subsequent questionnaires will be matched with the participant's data via their code number. Participants or their guardians will be required to remember their individual code, although, in the event they forget their code number, a master list will be kept on an external hard-drive in an encrypted, password-protected file, locked in the researchers' office.

During or shortly after the food-diary week, the researcher will schedule a meeting with each participant and guardian in order to provide detailed instructions on the first phase of the study and to obtain informed consent for continuation in the study from the parent/guardian and assent from the child. During the first meeting parents/guardians will complete study outcome measures. Child participants will also complete outcome measures and cognitive tests. These measures will be administered once again following the completion of the first phase (week five), following the four-week wash-out period (week nine), and the second phase (week thirteen). These measures are the clinical trial's primary end-points.

Following the information-gathering week, participants will begin the first phase of the study. They will consume either the probiotic or placebo powder taken with milk or ice cream for four weeks. For the second phase, the conditions will be reversed, and the participant will consume the alternate substance for four weeks; thus, all participants will receive the probiotic in one phase and the placebo in another phase. The order in which participants receive the probiotics and placebo will be randomized within groups of ten participants to ensure counterbalancing - i.e., roughly equal numbers of participants receiving probiotics and placebo in the first phase. The four-week intervention phases will be separated by a four-week washout period to ensure that any potential residual effects from the first phase have passed by the time the second phase commences. Following the wash-out period, participants will complete the relevant outcome measures once again to establish baseline scores prior to beginning the second intervention phase. Because this a double-blind design, the participants, their parents/guardians and the researchers administering the probiotics and placebos will not be aware which powder (probiotic or placebo) the participant is receiving in each of the two phases; only the Clinical Director at Lallemand Health Solutions will be privy to the experimental condition of the participants. Morning saliva samples for cortisol analysis will be collected from participants during weeks two (baseline visit), five (second visit), nine (third visit), and thirteen (fourth visit) of the study.

During the first week of each phase, the researcher will contact the participants by email or phone on the third and sixth day to check in and make sure participants/their guardians do not have any concerns and/or questions regarding their participation. Following the initial week of each phase, participants will be contacted weekly in order to monitor progress and address any concerns.

During first and second meetings, parents will be supplied with either probiotic or placebo powder as well as detailed instructions for the first and second intervention phases. At the fourth and final appointment, participants will complete the aforementioned questionnaires (if not done online) and be given the opportunity to ask any questions they may have about the study. If participants wish to know during which phase they received the probiotic formula, they be supplied with this information following the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* average score of 2.5 or higher on either the hyperactive/impulsive or inattentive symptoms on eligibility questionnaire
* total score of 10 or higher on the anxiety eligibility questionnaire

Exclusion Criteria:

* Dairy or Soy allergy
* Currently taking antibiotics
* HIV/AIDS
* Diagnosis of Cancer, Crohn's Disease, or Ulcerative Colitis
* Undergoing chemotherapy

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD-specific items of the Child Disruptive Behavior Disorders Scale | First day of study participation and again at weeks 4, 8, and 12

SECONDARY OUTCOMES:
Change in Salivary cortisol | First day of study participation and again at weeks 4, 8, and 12
Change in total score on the Screen for Child Anxiety Related Emotional Disorders | First day of study participation and again at weeks 4, 8, and 12
Change in Word Pairs Memory Test | First day of study participation and again at weeks 4, 8, and 12
Change in Visual Memory Test | First day of study participation and again at weeks 4, 8, and 12
Change in total omission and commission errors on the Continuous Performance Task | First day of study participation and again at weeks 4, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Susan Potter, Phd., Principal Investigator — Acadia University
Locations (1):
- Acadia University, Wolfville, Nova Scotia, Canada